CLINICAL TRIAL: NCT00177398
Title: The Effect of Insulin Glargine on Glycemic Control, Morbidity, and Length of Stay in Hospitalized Subjects With Diabetes Receiving Enteral Nutrition
Brief Title: Effect of Glargine Insulin on Glucose Control in Hospitalized Patients Who Receive Tube Feedings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB0408186
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Type 2 Diabetes; Hyperglycemia
Keywords: Type 2 diabetes; Hyperglycemia; Enteral nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

INTERVENTIONS:
Drug: Glargine insulin vs regular insulin

SUMMARY:
The purpose of this study is to determine if the early initiation of a long acting insulin (i.e. glargine) with supplemental doses of short acting regular (SSR) insulin in hospitalized patients with diabetes who are fed using tube feedings reduces the frequency of high and low blood sugar levels when compared to use of SSR insulin alone.

DETAILED DESCRIPTION:
Hyperglycemia is one of the most frequently encountered complications of enteral nutrition therapy in the hospital setting. However, there is no standardized approach directed towards the identification and management of patients who develop hyperglycemia while receiving enteral nutrition. The primary aim of the study is to determine if the early initiation of subcutaneous glargine insulin with supplemental doses of sliding scale human regular (SSR) insulin in hospitalized subjects with diabetes receiving enteral nutrition reduces the frequency of hyperglycemia and hypoglycemia when compared to use of SSR insulin alone.

In this proposal, we plan to investigate a strategy of early insulin therapy in the management of hospitalized subjects with diabetes mellitus who develop hyperglycemia defined as two blood glucose (BG) measurements greater than 130 mg/dl within 48 hours prior to or within a 48 hour period during enteral nutrition therapy.

The study is a phase IV, investigator initiated randomized, parallel group clinical trial. Potential subjects will include those subjects with written orders for initiation of enteral feedings using a formula containing carbohydrates. Consented subjects will have bedside glucose monitoring performed every 6 hours for the first 48 hours following initiation of enteral nutrition to determine if hyperglycemia occurs. To determine a difference in mean plasma glucose of 25 mg/dl and hospital LOS of 4 days between the two groups with an of 0.01 with power of 0.9, 25 subjects will be randomized to each group (total of 50 subjects). Baseline and outcome variables between the two groups will be compared using Student's t-testing, chi-square analysis, and the Mann-Whitney U test.

Group 1 will receiving a single daily dose of glargine insulin along with sliding scale regular human (SSR) insulin titrated according to blood glucose results. Group 2 will receive only sliding scale human regular (SSR) insulin titrated according to an algorithm. Both groups will be followed daily until enteral feedings are discontinued or for a maximum of three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes defined according to ADA criteria
* Enteral nutrition therapy
* Two blood glucose readings > 130 mg/dl within 48-hrs prior to or within a 48-hour period during enteral nutrition therapy
* Men and women age >/= 18
* Ability for patient or legally authorized representative to understand and sign an informed consent document

Exclusion Criteria:

* Subjects with conditions that are anticipated to have short term (i.e. < 2 months survival) based on discussions with the treatment team and attending physician.
* Subjects admitted to the CT ICU or any unit with pre-established protocols for glycemic management.
* Subjects with known type 1 diabetes (who will absolutely require a long or intermediate acting insulin preparation).
* Subjects with known type 2 diabetes who currently receive 30 units or more of an intermediate or long acting insulin.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-02; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome to be studied is the frequency and severity of hyperglycemia and hypoglycemia in each group
Time to mean 24 hour plasma glucose < 180 mg/dl

SECONDARY OUTCOMES:
Triglyceride level at study entry and conclusion
Hospital length of stay
Inpatient mortality
Number of days of antibiotic therapy
Number of days with recorded temperature >/= 100.4F
Occurrence of any of the following: MI, CHF, pneumonia, CVA, renal impairment (defined as serum creat > 2 mg/dl)
Quality of Life measures using MOS SF 36 General Health Survey
Outpatient glycemic control and self management practices

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Korytkowski, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Pancorbo-Hidalgo PL, Garcia-Fernandez FP, Ramirez-Perez C. Complications associated with enteral nutrition by nasogastric tube in an internal medicine unit. J Clin Nurs. 2001 Jul;10(4):482-90. doi: 10.1046/j.1365-2702.2001.00498.x. PMID 11822496
- [Background] Clement S, Braithwaite SS, Magee MF, Ahmann A, Smith EP, Schafer RG, Hirsch IB; American Diabetes Association Diabetes in Hospitals Writing Committee. Management of diabetes and hyperglycemia in hospitals. Diabetes Care. 2004 Feb;27(2):553-91. doi: 10.2337/diacare.27.2.553. No abstract available. PMID 14747243
- [Derived] Korytkowski MT, Salata RJ, Koerbel GL, Selzer F, Karslioglu E, Idriss AM, Lee KK, Moser AJ, Toledo FG. Insulin therapy and glycemic control in hospitalized patients with diabetes during enteral nutrition therapy: a randomized controlled clinical trial. Diabetes Care. 2009 Apr;32(4):594-6. doi: 10.2337/dc08-1436. PMID 19336639